CLINICAL TRIAL: NCT02996214
Title: A Multicenter, Randomized, Open-label, Parallel-group Study of Paclitaxel Liposome and Cisplatin Compared With Gemcitabine and Cisplatin as First-line Therapy in Advanced Squamous Non-Small-Cell Lung Cancer
Brief Title: Paclitaxel Liposome for Squamous Non-Small-cell Lung Cancer Study(LIPUSU)
Acronym: LIPUSU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing Luye Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY-TM-LPS-2016-01
Record Dates: First submitted 2016-12-04; First posted 2016-12-19 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Squamous Non-small-cell Lung Cancer
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LP group (Experimental): Liposome paclitaxel(Lipusu®) plus cisplatin. Paclitaxel liposome Sterile injection powder 175 mg/m^2, given on day 1 of a 21-day cycle, for 4-6 cycles. Cisplatin 75 mg/m^2, given on day 1 of a 21-day cycle, for 4-6 cycles.
  Interventions: Drug: Paclitaxel Liposome; Drug: Cisplatin
- GP group (Active Comparator): Gemcitabine (Gemzar®) plus cisplatin. Gemcitabine hydrochloride for injection 1000 mg/m^2, given on days 1 and 8 of a 21-day cycle, for 4-6 cycles. Cisplatin 75 mg/m^2, given on day 1 of a 21-day cycle, for 4-6 cycles.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel Liposome — Paclitaxel liposome injection 175 mg/m^2, given on day 1 of a 21-day cycle, for 4-6 cycles.
  Other Names: Lipusu®
  Arms: LP group
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2, given on days 1 and 8 of a 21-day cycle, for 4-6 cycles.
  Other Names: Gemzar®
  Arms: GP group
Drug: Cisplatin — Cisplatin 75 mg/m^2, given on day 1 of a 21-day cycle, for 4-6 cycles.
  Other Names: Nuoxin®

SUMMARY:
The purpose of this study is to investigate the efficacy and the safety of paclitaxel liposome and cisplatin compared with gemcitabine and cisplatin as first-line therapy in advanced squamous non-small-cell lung cancer .

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy and safety of paclitaxel liposome and cisplatin compared with gemcitabine and cisplatin as first-line therapy in advanced squamous non-small-cell lung cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old, both gender;
2. ECOG: 0-1;
3. Squamous non-small-cell lung cancer (stage IIIB or IV) confirmed by histologically or cytologically ;
4. No prior chemotherapy, biological therapy or immunotherapy; or subjects have recurrence and metastasis more than 6 months after the end of chemotherapy, but not gemcitabine or paclitaxel;
5. At least one radiographically measurable or assessable lesion on chest CG according to RECIST1.1 (response evaluation criteria of solid tumors); regional lymph node metastases may also be measured or assessed by imaging (mediastinal lymph nodes);
6. Life expectancy of at least 12 weeks;
7. Before treatment, blood tests or biochemical measurements must meet the following criteria:

   * White blood cell count (WBC)≥ 4.0*10^9/L;
   * Neutrophil count (ANC)≥ 2.0*10^9/L;
   * Platelet count (PLT)≥ 100*10^9/L;
   * Hemoglobin (Hb)≥ 100g/L;
   * Hepatic function: serum bilirubin ≤ 1.5 times the upper normal limit,aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper normal limit;
   * Renal function: creatinine ≤ 1.5 times the upper normal limit;
8. Signed informed consent.

Exclusion Criteria:

1. Hypersensitivity reaction to the interventional drugs;
2. Pregnant or breastfeeding;
3. Women or men of childbearing age who disagree with the use of effective contraceptive measures during the study period;
4. Brain metastase ;
5. Uncontrolled pleural effusion in patients with squamous non-small-cell lung cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From study entry to measured progressive disease, up to 2 years
  Progression free survival will be calculated from study entry to documented disease progression using RECISTv1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | From study entry to measured progressive disease, up to 2 years
  Objective response rate is the percentage of participants who achieve best overall tumor response of complete response or partial response .
Overall Survival | From study entry to death from any cause, up to 2 years
  Overall survival is defined from study entry to the date of death from any cause.
Adverse events | From baseline until 21 days after the last dose
  Adverse events is evaluated according to Common Terminology Criteria for Adverse Events Version 4.0
Quality of Life questionnaire | From study entry to measured progressive disease, up to 2 years
  The quality of life is assessed using the European Organization for the Research and Treatment of Cancer Questionnaire Core-30 (EORTC QLQ-C30) and Quality of Life Questionnaire Lung Cancer 13(QLQ-LC13).
Correlation between gene sequence or expression level and therapeutic effect | From study entry untill radiological disease progression, up to 2 years
  Correlation between gene sequence or expression level and therapeutic effect is assessed using the blood or tumor tissue of subjects by genetic testing

CONTACTS AND LOCATIONS:
Overall Officials: caicun zhou, doctor, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Pan Y, Shi Q, Zhang G, Jiang L, Dong X, Gu K, Wang H, Zhang X, Yang N, Li Y, Xiong J, Yi T, Peng M, Song Y, Fan Y, Cui J, Chen G, Tan W, Zang A, Guo Q, Zhao G, Wang Z, He J, Yao W, Wu X, Chen K, Hu X, Hu C, Yue L, Jiang D, Wang G, Liu J, Yu G, Li J, Bai J, Xie W, Zhao W, Wu L, Zhou C. Paclitaxel liposome for injection (Lipusu) plus cisplatin versus gemcitabine plus cisplatin in the first-line treatment of locally advanced or metastatic lung squamous cell carcinoma: A multicenter, randomized, open-label, parallel controlled clinical study. Cancer Commun (Lond). 2022 Jan;42(1):3-16. doi: 10.1002/cac2.12225. Epub 2021 Oct 26. PMID 34699693